CLINICAL TRIAL: NCT06091852
Title: The Incorporation of Dietary Protein-Derived Amino Acids in Duodenal Mucosal Protein in Young and Older Males
Brief Title: The Incorporation of Dietary Protein-Derived Amino Acids in Duodenal Epithelium
Acronym: GutFeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: METC23-011
Record Dates: First submitted 2023-06-27; First posted 2023-10-19 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2023-10

CONDITIONS: Protein Malabsorption
Keywords: Gastrointestinal tract; Intestinal mucosa; Protein; Digestion; Absorption; Aging; Muscle protein synthesis

STUDY DESIGN:
Intervention Model Description: Young vs. old
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intrinsically labelled milk protein (Experimental): 20 grams of protein dissolved in 500 mL of water
  Interventions: Dietary Supplement: Intrinsically labelled milk protein

INTERVENTIONS:
Dietary Supplement: Intrinsically labelled milk protein — 20 grams of protein dissolved in 500 mL of water

SUMMARY:
Rationale: Aging is accompanied by a blunted muscle protein synthetic response to protein ingestion.This anabolic resistance may be related to decreased postprandial amino acid release in the circulation, due to greater amino acid extraction by splanchnic tissues in older individuals. It has been suggested that extracted amino acids are utilized by intestinal epithelial cells for cell proliferation, generating new cells to maintain healthy mucosa. So far, there is no evidence that dietary protein-derived amino acids are taken up and incorporated in intestinal mucosal protein in vivo in humans. Furthermore, there is no evidence that this process is impacted by age.

Objective: To assess the postprandial incorporation of dietary protein-derived amino acids in intestinal mucosal protein in healthy young and older males.

Study design: Cross-sectional, non-therapeutic intervention study design

Study population: 5 healthy, non-obese (BMI 18.5-30kg/m2) young adult males (age: 18-35y inclusive) and 5 community dwelling older males (age: 67+y).

Intervention: Continuous intravenous stable isotope amino acid tracer infusion will be applied, in combination with oral ingestion of 20g intrinsically labelled milk protein, with plasma, muscle and duodenal mucosa biopsy samples collected at different time points throughout the experimental test day.

Main study parameters/endpoints: The primary study outcome is the postprandial (0-5h) incorporation of dietary protein-derived amino acids in duodenal mucosal protein following the ingestion of 20g intrinsically labelled milk protein. Secondary study parameters include postprandial plasma availability of dietary protein-derived amino acids and fractional duodenal mucosal protein synthetic rate.

DETAILED DESCRIPTION:
Skeletal muscle tissue is in a constant state of remodelling, regulated by the balance between tissue protein synthesis and breakdown rates, with a turnover rate of 1-2% per day. It has been well established that protein ingestion is a major anabolic stimulus for muscle protein synthesis. Dietary protein ingestion provides amino acids that stimulate protein synthesis by both functioning as substrate and as signalling molecules that upregulate anabolic pathways.

The anabolic properties of dietary protein largely depend on the protein digestion and amino acid absorption kinetics and subsequent increase in plasma amino acid availability. Following protein ingestion, protein is cleaved into small peptides and amino acids by digestive enzymes. Subsequently, these amino acids are absorbed across the intestinal mucosa by various membrane-bound transporters. The majority of dietary protein derived amino acids is released into the systemic circulation and transported and taken up by various peripheral tissues in the postprandial phase. However, a substantial part of the ingested protein does not become available in the circulation. This part is either not (yet) digested and absorbed, or the absorbed amino acids are taken up by splanchnic tissues, such as the gut and liver, providing precursors for de novo tissue protein synthesis, termed first-pass splanchnic extraction. Previous work in our laboratory has estimated that up to 40% of the protein derived amino acids are taken up and incorporated in the intestinal tract and liver tissues. The intestine is the most highly regenerative organ in the human body, regenerating its epithelium every 3 to 5 days. It has been suggested that the absorbed amino acids are utilized by epithelial cells for rapid cell proliferation, generating new cells to maintain healthy mucosa. Human studies on the incorporation of dietary protein-derived amino acids in intestinal mucosal protein have not been performed. Therefore, the aim of the present explorative in vivo study is to assess, for the first time, the incorporation of dietary protein-derived amino acids in duodenal mucosal protein in humans, and the systemic availability of dietary protein-derived amino acids.

Aging is accompanied by a blunted muscle protein synthetic response to protein ingestion. This proposed anabolic resistance may be related to a decreased postprandial amino acid release in the circulation, due to impairments in protein digestion and amino acid absorption, and greater first-pass splanchnic amino acid extraction in older individuals. Whether dietary protein-derived amino acid incorporation in intestinal mucosal protein is increased with aging remains to be established. Therefore, the current study will use the data on incorporation of dietary protein-derived amino acids in duodenal mucosal protein and postprandial amino acid plasma availability obtained in young and older individuals to evaluate potential age-related differences.

Two primary hypotheses will be tested:

1. It is hypothesized that part of the absorbed amino acids will be directly incorporated in duodenal epithelium within 5 hours after protein ingestion.
2. It is hypothesized that the extent of postprandial incorporation of dietary protein derived amino acids in duodenal epithelium will be greater in older compared to young males.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Aged 18-35 years or 67+ years
* Body mass index (BMI) between 18.5 and 30 kg/m2

Exclusion Criteria:

* History of cardiovascular, respiratory, gastrointestinal, urogenital, neurological, psychiatric, dermatologic, musculoskeletal, metabolic, endocrine, haematological, immunologic disorders, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol, interfere with the execution of the experiment, or potential influence the study outcomes (to be decided by the principal investigator and responsible physician)
* Major abdominal surgery interfering with gastrointestinal function (upon judgement of the principal investigator and responsible physician)
* Use of medication which limit participation in or completion of the study protocol, interferes with the execution of the experiment, or potential influences the study outcomes (to be decided by the principal investigator and responsible physician)
* Use of supplementation (i.e. vitamin, pre- and probiotic supplementation) within 14 days prior to testing
* Administration of investigational drugs or participation in any scientific intervention study in the 14 days prior to the study, which may interfere with this study (upon judgement of the principal investigator and responsible physician)
* Specific diet (e.g. vegetarian, vegan, gluten free, no diary) within the study period
* Planning to lose weight during the study period
* Lactose intolerance
* Excessive alcohol consumption (defined as > 14 alcoholic consumptions per week)
* Smoking
* Drug use
* Donated blood two months prior to the test day
* Recent (<1 year) participation in amino acid tracer (L-[ring-2H5]-phenylalanine, L-[ring-2H3]-leucine, L-[ring-2H4]-lysine, L-[ring-2H2]-tyrosine) or intrinsically labelled protein ([1-13C]-phenylalanine, [1-13C]-leucine, [1-13C]-lysine) studies
* No given permission to register participation in electronic patient file at MUMC+ and to add records of gastroduodenoscopy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

PRIMARY OUTCOMES:
Postprandial incorporation of dietary protein-derived amino acids in duodenal mucosal protein | 0-5 hours
  Assessed by duodenal mucosal protein-bound [1-13C]-phenylalanine enrichment (expressed as MPE)
Impact of age on postprandial incorporation of dietary protein-derived amino acids in duodenal mucosal protein | 0-5 hours
  Assessed by duodenal mucosal protein-bound [1-13C]-phenylalanine enrichment (expressed as MPE) in young and older adults

SECONDARY OUTCOMES:
Postprandial plasma amino acid concentrations | 0-5 hours
  Appearance of milk protein-derived amino acids in plasma over the full assessment period (5 h), as determined using stable isotope tracer methodology
Fractional duodenal mucosal protein synthetic rate | 0-5 hours
  Mucosal protein synthesis rates are calculated using L-ring-2H5-phenylalanine tracer and provided as 1 integrated value over the specified timeframe using plasma as precursor
Fractional muscle protein synthetic rate | 0-5 hours
  Muscle protein synthesis rates are calculated using L-ring-2H5-phenylalanine tracer and provided as 1 integrated value over the specified timeframe using plasma as precursor
Fecal [1-13C]-phenylalanine enrichments (expressed as MPE) | Fecal sample of first feces after endoscopy
  Fecal protein excretion, assessed by fecal [1-13C]-phenylalanine enrichments (expressed as MPE)
Fecal nitrogen content | Fecal sample of first feces after endoscopy
  Fecal protein excretion, assessed by fecal nitrogen content
Fecal microbial metabolites | Fecal sample of first feces after endoscopy
  Microbial metabolites, including short-chain fatty acids, assessed by analyzing fecal samples
Plasma glucose concentrations | 0-5 hours
  Plasma glucose concentrations
Plasma insulin concentrations | 0-5 hours
  Plasma insulin concentrations

OTHER OUTCOMES:
Age in years | Baseline
  Reported by participants
Body weight in kg | Baseline
  Scale
Height in m | Baseline
  Stadiometer
BMI in kg/m2 | Baseline
  Calculated from height and body weight
Skeletal muscle mass | Baseline
  Bioelectrical impedance analysis
Fat mass | Baseline
  Bioelectrical impedance analysis
Dietary macronutrient intake | 2 days prior to experimental trial day
  Assessed by written dietary intake records
Systolic blood pressure in mmHg | Baseline
  Electrical sphygmomanometer
Diastolic blood pressure in mmHg | Baseline
  Electrical sphygmomanometer

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, Prof, Principal Investigator — Maastricht University Medical Center; Daisy Jonkers, Prof, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No